CLINICAL TRIAL: NCT06833333
Title: Role of Inferior Vena Cava Collapsibility Index or Central Venous Pressure as a Predictor of Fluid Responsiveness in Pediatric Sepsis Due to Perforated Viscus: Prospective Randomized Double-blind Study
Brief Title: IVC Collapsibility Index or CVP as a Predictor of Fluid Responsiveness in Pediatric Sepsis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1033/1/25
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Sepsis; Septic Shock; Perforated Viscus; Hospitalism in Children
Keywords: Pediatric; sepsis; Fluid therapy
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Central Venous Catheters

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigated patients are children aged 1-5 years. Measurements will be obtained by an assistant nurse not participating in the study and blinded to its groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (CVP) (Experimental): patients in this group will receive fluid resuscitation and therapy guided by central venous pressure.
  Interventions: Procedure: Central venous catheter
- Group II (IVC) (Experimental): patients in this group will receive fluid resuscitation and therapy guided by IVC collapsibility index.
  Interventions: Procedure: Central venous catheter; Diagnostic Test: IVC collapsibility index

INTERVENTIONS:
Procedure: Central venous catheter — Central venous catheter will be introduced to measure central venous pressure
Diagnostic Test: IVC collapsibility index — In supine position, IVC will be assessed in the anteroposterior plane in the subxiphoid view using two-dimensional mode till an optimal view of IVC entering the right atrium will be obtained. Then, measurement of its collapsibility will be done.
  Arms: Group II (IVC)

SUMMARY:
Pediatric population who suffered from sepsis due to perforated viscus will receive fluid resuscitation guided by either central venous pressure or guided by IVC collapsibility index.

The method of guidance of fluid therapy will be applied pre, intra, and postoperatively.

Primary outcome will be the length of hospital stays, while the secondary outcomes will be the incidence of complications and the length of PICU stays

DETAILED DESCRIPTION:
This prospective randomized double-blind study will be carried out on 44 pediatric patients who will be presented to Tanta university hospitals with sepsis owing to perforated viscus, an informed written consent will be obtained from all the parents of the participants, all patients data will be confidential and will be used for the current study only.

Ethical Considerations

Pediatric patients aged 1 to 5 years presented with septic shock due to perforated viscus according to definition of the American College of Critical Care Medicine and International Pediatric Sepsis Consensus will be included

Patients will be randomly classified using a computer-generated software of randomization into 2 groups:

Group I (CVP group): patients in this group will receive fluid resuscitation and therapy guided by central venous pressure.

Group II (IVC group): patients in this group will receive fluid resuscitation and therapy guided by IVC collapsibility.

Patient management Pediatric patients presented with septic shock will be admitted to pediatric intensive care unit (PICU). Intravascular access was established with starting mechanical ventilation and resuscitation. Fluid resuscitation in the form of 10 ml/kg of lactated ringer over 10 minutes will be started if there is one or more of the followings; a) severe tachycardia, b) decrease in systolic blood pressure, c) decrease in urine output less than < 0.5 mL/kg/h, d) prolongation of capillary refill time more than 5 seconds. An ultrasound-guided central venous catheter will be applied. Blood samples will be obtained to measure complete blood count, the renal function, coagulation studies, plasma electrolytes, C- reactive protein, and arterial blood gases. Plain erect X-ray will be done to all patients together with pelvi-abdominal ultrasound.

After initial fluid resuscitation, the fluid therapy volume will be directed according to either central venous pressure or IVC collapsibility index. In group I, the CVP will be measured after initial fluid resuscitation and lactated ringer solution 2 ml/kg over 20 minutes will be given intravenously and can be repeated until reaching CVP of more than 8 mmHg or reaching a total volume of ringer solution to 20 ml/kg. Failure to obtain adequate CVP either maximal dose of fluid (20 ml/kg) or failure to obtain adequate hemodynamics after fluid therapy will be managed by starting vasopressor therapy or inotropic therapy.

In the second group, ultrasound-guided IVC collapsibility index will be done after initial fluid bolus therapy. Lactated ringer solution 2 ml/kg over 20 minutes that can be repeated will be given and repeated until reaching IVC collapsibility index less than 30 % or reaching maximal dose of fluid (20 ml/kg). vasopressor and inotropic therapy will be started if the IVC collapsibility index is not reached despite reaching maximal fluid dose or in failure to obtain stable hemodynamics despite maximal fluid resuscitation.

Once the child is stabilized, he will be admitted to the operating room and received general anesthesia and connected to 5 ASA basal monitors (pulse oximeter, 5-leads ECG, non-invasive blood pressure, End-tidal carbon dioxide, and temperature). The intraoperative fluid and vasopressor therapy will be directed by either CVP or IVC collapsibility index according to the patient group. After completing the surgery, the child will be transported to the PICU on mechanical ventilator with postoperative fluid and vasopressor management according to CVP or IVC collapsibility index according to the patient group. The child general condition, daily laboratory investigations, arterial blood gases, and incidence of complications will be monitored closely.

Measurements:

Primary outcome will be the length of hospital stays, while the secondary outcomes will be the incidence of complications and the length of PICU stays

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 1 to 5 years presented with septic shock due to perforated viscus according to definition of the American College of Critical Care Medicine and International Pediatric Sepsis Consensus.

Exclusion Criteria:

* Refusal of the parents to participate in the study
* Obesity
* Congenital heart diseases
* Severe arrythmias
* Patients developed moderate to severe ARDS
* Massive ascites
* Previous abdominal surgery
* Previous cardiothoracic surgery

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
the length of hospital stays | within first 28 days
  The number of days from admission of the child till discharge

SECONDARY OUTCOMES:
The length of PICU stays | within first 28 days
  The number of days from admission of child to ICU till discharge from ICU.
The incidence of complications | within first 28 days
  The incidence of acute kidney injury, ARDs, acidosis, severe oedema, or mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Once the study had been successfully completed, the data will be shared for other researchers
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months from publication of the study